CLINICAL TRIAL: NCT02106949
Title: Short Message System (SMS) Monitoring Intended for the Suicidal Patients: Study of Efficiency
Brief Title: Short Message System (SMS) Monitoring Intended for the Suicidal Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Technopôle Brest-Iroise: LANESTEL SARL, 38 rue Jim Sevellec, 29200 Brest (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SIAM; RB 13-068 [CHRU Brest]
Record Dates: First submitted 2014-04-04; First posted 2014-04-08 (Estimated); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Patients Having Realized a Suicide Attempt
Keywords: suicide attempt, SMS monitoring, recurrence, phone, prevention control, tertiary healthcare
MeSH Terms: conditions — Suicide, Attempted; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS (Experimental): The patients of the test group receive a first SMS 48 hours after their discharge from the hospital then a total of 10 messages distributed over six months: 48 hours, S1, S2, M1, M2, M3, M4, M5, M6 and M13.
  Interventions: Device: SMS contact with patient after discharge in intervention group
- Without SMS (No Intervention): The patients of the group benefit from the usual care.

INTERVENTIONS:
Device: SMS contact with patient after discharge in intervention group
  Arms: SMS

SUMMARY:
The study wants to prove that SMS monitoring reduced the number of suicide attempts in six months according to the beginning of its implementation in the group of the patients benefiting SMS compared with the group of patients benefiting from the usual care.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Surviving a suicide attempt
* Leaving directly the emergency department or hospitalized less than 7 days
* Being able to be joined by telephone mobile

Exclusion Criteria:

* under guardianship
* Patient who are not able to provide a consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2014-08-20 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

PRIMARY OUTCOMES:
Number of suicide reattempts in every group | 6 months

SECONDARY OUTCOMES:
Number of suicide reattempts in every group | 13 months
Total number of suicidal second recurrences in every group | 6 months
Total number of suicidal second recurrences in every group | 13 months
Number of deaths by suicide | 6 months and 13 months
Score in the scale C-SSRS | inclusion, 6 months and 13 months
Presence of a disorder in the MINI: characterization of the comorbidity | 6 months and 13 months

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU Angers, Angers
  - CHRU de Brest, Brest
  - CHU Caen, Caen
  - CHRU Lille, Lille
  - CHU de Lyon, Lyon
  - CHU Nantes, Nantes
  - CH Quimperlé, Quimperlé
  - CHU Rennes, Rennes
  - CHU de Saint-Etienne, Hôpital Nord, Saint-Etienne
  - CHU St Nazaire, Saint-Nazaire
  - CH St Malo, St-Malo
  - CHU Tours, Tours
  - CH Vannes, Vannes

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- [Derived] Berrouiguet S, Larsen ME, Mesmeur C, Gravey M, Billot R, Walter M; HUGOPSY Network; Lemey C, Lenca P. Toward mHealth Brief Contact Interventions in Suicide Prevention: Case Series From the Suicide Intervention Assisted by Messages (SIAM) Randomized Controlled Trial. JMIR Mhealth Uhealth. 2018 Jan 10;6(1):e8. doi: 10.2196/mhealth.7780. PMID 29321126
- [Derived] Berrouiguet S, Alavi Z, Vaiva G, Courtet P, Baca-Garcia E, Vidailhet P, Gravey M, Guillodo E, Brandt S, Walter M. SIAM (Suicide intervention assisted by messages): the development of a post-acute crisis text messaging outreach for suicide prevention. BMC Psychiatry. 2014 Nov 18;14:294. doi: 10.1186/s12888-014-0294-8. PMID 25404215